CLINICAL TRIAL: NCT01189448
Title: Multicenter, Randomized Clinical Trial to Compare the Efficacy and Tolerance of Prenatal Therapy With Pyrimethamine + Sulfadiazine vs Spiramycine to Reduce Vertical Transmission of Toxoplasma Gondii Following Primary Infection in Pregnancy
Brief Title: Prevention of Congenital Toxoplasmosis With Pyrimethamine + Sulfadiazine Versus Spiramycine During Pregnancy
Acronym: TOXOGEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081234; 2010-019972-65 (EudraCT Number)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Congenital Toxoplasmosis
Keywords: Congenital Toxoplasmosis,; Pregnancy,; prenatal diagnosis,; mother-to-child transmission,; prevention,; spiramycine,; pyrimethamine-sulfadiazine
MeSH Terms: conditions — Toxoplasmosis, Congenital | interventions — Pyrimethamine; Sulfadiazine; Spiramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyrimethamine/Sulfadiazine (Active Comparator): Women who are enrolled and randomised in Pyrimethamine + sulfadiazine group : Pyrimethamine 50 mg once daily orally and sulfadiazine 1g tid. orally, with supplemental folinic acid 50 mg once a week.
  Interventions: Drug: Pyrimethamine/Sulfadiazine
- Spiramycine (Active Comparator): Spiramycin group : spiramycin 1g tid orally
  Interventions: Drug: Spiramycine

INTERVENTIONS:
Drug: Pyrimethamine/Sulfadiazine — Pyrimethamine + sulfadiazine group : Pyrimethamine 50 mg once daily orally and sulfadiazine 1g tid. orally, with supplemental folinic acid 50 mg once a week.
  Follow-up includes clinical and biological tolerance, according to usual recommendations. Monthly fetal ultrasound is performed. Prenatal diagnosis with amniocentesis is offered after 18 weeks gestation, usually 4 weeks after the maternal infection.
  Treatment is be stopped or changed in case of toxicity. If prenatal diagnosis shows fetal infection with T. gondii, management is to be determined by the clinicians with the patient. If the prenatal diagnosis is negative the treatment can be stopped in order to reduce the risk of intolerance, providing that the mother receives at least 4 weeks of therapy.
  Other Names: Pyrimethamine = Malocide®; Sulfadiazine = Adiazine®
  Arms: Pyrimethamine/Sulfadiazine
Drug: Spiramycine — Spiramycin group : spiramycin 1g tid orally Follow-up includes clinical and biological tolerance, according to usual recommendations. Monthly fetal ultrasound is performed. Prenatal diagnosis with amniocentesis is offered after 18 weeks gestation, usually 4 weeks after the maternal infection.
  Treatment is be stopped or changed in case of toxicity. If prenatal diagnosis shows fetal infection with T. gondii, management is to be determined by the clinicians with the patient. If the prenatal diagnosis is negative the treatment is continued according to usual procedures
  Other Names: Spiramycine = Rovamycine®
  Arms: Spiramycine

SUMMARY:
Background : When a mother contracts toxoplasmosis during pregnancy, the parasite may be transmitted from to her unborn child. This results in congenital toxoplasmosis, which may cause damage to the eyes and nervous system of the child. To date, no method has been proved effective to prevent this transmission. In France, spiramycin is usually prescribed to women who have toxoplasma seroconversion in pregnancy, however its efficacy has not been determined. The standard treatment for toxoplasmosis is the combination of the antiparasitic drugs pyrimethamine and sulfadiazine, but this strategy has not been evaluated for the prevention of mother-to-child transmission.

Purpose : Randomized phase 3 trial to determine whether pyrimethamine + sulfadiazine is more effective than spiramycin to prevent congenital toxoplasmosis.

DETAILED DESCRIPTION:
The protocol is a comparison of 2 strategies to prevent mother-to-child transmission of T. gondii following maternal seroconversion.

Screening for toxoplasmosis is mandatory in France. Patients with confirmed seroconversion will be eligible for the trial, after 14 weeks gestational age.

Participants will be randomly allocated to one of the treatment groups, and will receive open-label pyrimethamine + sulfadiazine or spiramycin.

The protocol will not change the usual procedures for prenatal diagnosis, nor will it change the management of infected fetuses and neonates.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Toxoplasmosis infection acquired during the pregnancy documented by at least one negative serology in the first trimester and seroconversion with presence of specific IgG antibodies
* Gestational age > 14 weeks from last menstrual period
* Signature of informed consent

Exclusion Criteria:

* Lack of a documented negative serology during the pregnancy
* Antiparasitic therapy with spiramycin, pyrimethamine or sulfa drugs for more than 10 days after seroconversion and before randomization,
* Known allergy to any of the study drugs, serious allergic conditions or G6PD deficiency,
* Known hepatic or renal insufficiency,
* Other ongoing severe conditions in mother or fetus
* Lack of public health insurance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Rate of mother-to-child transmission | Up to six months after birth
  Rate of mother-to-child transmission of toxoplasma gondii, determined by PCR on amniocentesis and/or synthesis of specific antibodies by the neonate

SECONDARY OUTCOMES:
Secondary Outcome Measure | Up to six months after birth
  * Mother-to-child transmission rate according to the time between primary infection and start of therapy
  * Tolerance in mothers and neonates (grade 3-4 toxicities)
  * Severity of infection at birth in case of congenital toxoplasmosis (parasite load in amniotic fluid, clinical and biological signs)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mandelbrot, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Colombes, Hauts-de-Saine, France

IPD SHARING:
Plan to Share IPD: Undecided